CLINICAL TRIAL: NCT01958489
Title: Effect of Evacetrapib on the Pharmacokinetics of Pravastatin in Healthy Japanese and Non-Japanese Subjects
Brief Title: A Study of Evacetrapib in Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14625; I1V-MC-EIAW (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pravastatin (Experimental): Single 40 milligram (mg) oral dose of pravastatin administered on Day 1.
  Interventions: Drug: Pravastatin
- Evacetrapib + Pravastatin (Experimental): Oral doses of 130 mg evacetrapib administered once daily on Days 2 through 11, with a single oral dose of 40 mg pravastatin coadministered on Day 11.
  Interventions: Drug: Evacetrapib; Drug: Pravastatin

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
  Arms: Evacetrapib + Pravastatin
Drug: Pravastatin — Administered orally

SUMMARY:
The main purpose of this study is to look at the effect of evacetrapib on pravastatin levels in the blood when both drugs are taken at the same time. The study will also assess how well the body handles evacetrapib and pravastatin when given at the same time.

This study has two periods in fixed order. Each participant will enroll in both periods. This study will last approximately 25 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants, as determined by medical history and physical examination
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m²)
* Japanese participants must be first generation Japanese

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were administered 40 milligrams (mg) Pravastatin on Day 1 (Period 1) and 130 mg Evacetrapib on Days 2 through 11 and 40 mg Pravastatin coadministered on Day 11 (Period 2).
Groups:
- Pravastatin: 40 mg oral dose of pravastatin was administered on Day 1.
- Evacetrapib + Pravastatin: 130 mg oral dose of evacetrapib was administered once daily (QD) on Days 2 through 11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
Period: Period 1
Arm/Group | Pravastatin | Evacetrapib + Pravastatin
Started | 24 | 0
Received at Least 1 Dose of Study Drug | 24 | 0
Completed | 24 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Pravastatin | Evacetrapib + Pravastatin
Started | 0 (Participants who completed Period 1 treatment crossed over to Period 2 treatment) | 24 (Participants who started Period 2 treatment crossed over from Period 1 treatment)
Received at Least 1 Dose of Study Drug | 0 | 24
Completed | 0 | 23
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Pravastatin and Evacetrapib + Pravastatin: 40 mg oral dose of pravastatin was administered on Day 1. One hundred and thirty (130) mg oral dose of evacetrapib was administered QD on Days 2 through 11 and 40 mg oral dose of pravastatin was co-administered on Day 11.
Arm/Group | Pravastatin and Evacetrapib + Pravastatin
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Pravastatin
Time Frame: Day 1 and Day 11: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours postdose
Population: All participants who had evaluable Cmax results at the specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Pravastatin (Period 1): 40 mg oral dose of pravastatin was administered on Day 1.
- Evacetrapib + Pravastatin (Period 2): 130 mg oral dose of evacetrapib was administered QD on Days 2 through 11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
Arm/Group | Pravastatin (Period 1) | Evacetrapib + Pravastatin (Period 2)
Number analyzed (Participants) | 23 | 23
nanograms/milliliter (ng/mL) | 142 (31) | 128 (43)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of Pravastatin
Time Frame: Day 1 and Day 11: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours postdose
Population: All participants who had evaluable AUC(0-∞) at the specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliters (ng*h/mL)
Groups:
- Evacetrapib + Pravastatin (Period 2): 130 mg oral dose of evacetrapib was administered QD on Days 2 through11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
Arm/Group | Pravastatin (Period 1) | Evacetrapib + Pravastatin (Period 2)
Number analyzed (Participants) | 23 | 23
nanograms*hours/milliliters (ng*h/mL) | 257 (27) | 229 (37)

3. Primary Outcome: PK: Time of Maximum Observed Concentration (Tmax) of Pravastatin
Time Frame: Day 1 and Day 11: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours postdose
Population: All enrolled participants with evaluable tmax results at the specific time points.
Measure: Median (Full Range); unit: hours
Arm/Group | Pravastatin (Period 1) | Evacetrapib + Pravastatin (Period 2)
Number analyzed (Participants) | 23 | 23
hours | 1.00 [0.50 to 2.00] | 0.75 [0.50 to 1.50]

ADVERSE EVENTS:
Groups:
- 40 mg Pravastatin Japanese; 40 mg Pravastatin Non-Japanese: 40 mg oral dose of pravastatin was administered on Day 1.
- 130 mg Evacetrapib Japanese; 130 mg Evacetrapib Non-Japanese: 130 mg oral dose of evacetrapib was administered QD on Days 2 through 11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
- 40 mg Pravastatin + 130 mg Evacetrapib Japanese: 40 mg oral dose of pravastatin was administered on Day 1. 130 mg oral dose of evacetrapib was administered QD on Days 2 through11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
- 40 mg Pravastatin + 130-mg Evacetrapib Non-Japanese: 40 mg oral dose of pravastatin was administered on Day 1. 130 mg oral dose of evacetrapib was administered QD on Days 2 through 11 and a 40 mg oral dose of pravastatin coadministered on Day 11.
Arm/Group | 40 mg Pravastatin Japanese | 130 mg Evacetrapib Japanese | 40 mg Pravastatin + 130 mg Evacetrapib Japanese | 40 mg Pravastatin Non-Japanese | 130 mg Evacetrapib Non-Japanese | 40 mg Pravastatin + 130-mg Evacetrapib Non-Japanese
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 2/10 | 6/10 | 4/10 | 4/14 | 4/14 | 6/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg Pravastatin Japanese (N=10) | 130 mg Evacetrapib Japanese (N=10) | 40 mg Pravastatin + 130 mg Evacetrapib Japanese (N=10) | 40 mg Pravastatin Non-Japanese (N=14) | 130 mg Evacetrapib Non-Japanese (N=14) | 40 mg Pravastatin + 130-mg Evacetrapib Non-Japanese (N=13)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.